CLINICAL TRIAL: NCT00579631
Title: Health Behaviors in Adolescent Survivors of Cancer or Similar Illnesses
Brief Title: Adolescent Survivors of Cancer or Similar Illnesses
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-074
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Adolescent Cancer Survivors; Pediatric Cancer Survivors
Keywords: survivors; adolescent; pediatric
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Questionnaire or Interview
  Interventions: Behavioral: Questionnaire or Interview

INTERVENTIONS:
Behavioral: Questionnaire or Interview — Complete a self-report survey once over the telephone or by mail. The questions are about your health beliefs and behaviors, your current health, and your mood. It should not take longer than 45 minutes to complete. About 15 of these people will participate in an additional, short audiotaped interview about sun protection.

SUMMARY:
The purpose of this study is to examine the health behaviors of young adults who have been treated for cancer, leukemia, or similar illnesses. We will also ask you some questions about your family members' and friends' health behaviors. We plan to use the findings from this study to design new programs to help teenage cancer survivors resist doing things that might harm their health.

DETAILED DESCRIPTION:
This study proposes to explore cancer-risk behaviors and future behavioral intentions among adolescent cancer survivors (i.e., 14-19 years old) and compare them to their "healthy" peers using population-based normative data. Additionally, it seeks to determine the significant theory-driven covariates related to adolescent survivors' health behaviors, which will aid in the design of future behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

* Current age at enrollment between 14 and 19;
* A diagnosis of cancer between the ages of 8 and 14;
* At least 12 months post-treatment and no evidence of disease (NED) at the time of assessment;
* Can be reached by mail or telephone;
* Fluent in English;
* Parent or legal guardian able to provide informed consent;
* Able to provide informed assent.

Exclusion Criteria:

* Major psychopathology or cognitive impairment likely in the judgment of the investigator to interfere with participation and compliance with the protocol.
* Currently receiving therapy for cancer treatment

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Memorial Sloan-Kettering Cancer Center's Department of Pediatrics
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2004-06-22 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
To describe the patterns of cancer-risk behaviors for adolescent cancer survivors as compared to population-based normative data of "healthy" adolescents, and to describe relevant theory-driven covariates for adolescent cancer survivors. | conclusion of study

SECONDARY OUTCOMES:
To examine the role and relative utility of sociodemographics, medical characteristics, theory-driven variables in explaining adolescent cancer survivors' health behaviors. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Marie Barnett, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org